CLINICAL TRIAL: NCT07293455
Title: Evaluation and Demonstration of New Tuberculosis Diagnostics for Indonesia; Work Package 3: Cluster Randomised Controlled Trial of A Diagnostic Package to Increase the Number of Tuberculosis Cases Notified
Brief Title: Evaluation and Demonstration of New Tuberculosis Diagnostics for Indonesia
Acronym: EVIDENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Otago (Other); University of Melbourne (Other); Radboud University Medical Center (Other); Universitas Sebelas Maret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TBWG-202511.01
Record Dates: First submitted 2025-12-05; First posted 2025-12-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Diagnosis; Tongue swab; Near point-of-care test; Cluster randomised controlled trial
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statisticians and investigators who will conduct the primary data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near Point-of-Care (nPOC) Testing (Active Comparator): The intervention arm will comprise HCFs operating in the selected CHC catchment areas, including CHCs, public hospitals, private hospitals, private clinics, and private laboratories. A multi-component public health intervention package, which will incorporate nPOC testing for TB diagnosis, will be provided for these HCFs, including patients visiting the HCFs and the community residents in the selected CHC catchment areas.
  Interventions: Diagnostic Test: nPOC Testing Intervention Package
- Standard of Care (No Intervention): HCFs in the control arm will continue standard of care with no intervention, except for refresher training on reporting and notifying TB cases to the National TB Information System before the intervention package is rolled out.

INTERVENTIONS:
Diagnostic Test: nPOC Testing Intervention Package — The intervention package will comprise:
  1. Introduction of a new-generation diagnostic test (nPOC test) into the HCFs;
  2. Optimisation of clinical algorithms with the incorporation of the new test;
  3. Promotional package to encourage patient attendance and utilisation of tests at HCFs by practitioners in the intervention areas;
  4. TB household contact investigation using the new test according to an algorithm with community health volunteers (cadres) involvement in the intervention areas.
  Arms: Near Point-of-Care (nPOC) Testing

SUMMARY:
The goal of this cluster-randomised controlled trial (CRCT) is to learn whether the use of new non-sputum-based diagnostic tests and other intervention components for tuberculosis (TB) diagnosis in healthcare facilities (HCF) can increase TB notifications. The main questions it aims to answer are: (1) Does the diagnostic intervention package raise TB notifications by HCF?; (2) Does the diagnostic intervention package raise the proportion of patients with TB who are diagnosed with microbiological tests, lower the time needed for TB diagnosis, lower the number of visits to HCF before TB diagnosis, raise the use of TB tests by healthcare providers, and lower the costs for TB diagnosis?

Researchers will compare the diagnostic intervention package provided to HCFs and the community in the intervention arm with the standard of care in the control arm to assess the intervention's effect. Healthcare providers will be trained to provide diagnostic interventions to patients visiting their HCFs and to community residents in the areas surrounding HCFs.

DETAILED DESCRIPTION:
TB remains a critical public health problem worldwide. Most of the patients with TB were from low- and middle-income countries with limited resources. A large proportion of them visited HCFs without sufficient laboratory services to diagnose TB, causing a delay in TB diagnosis and treatment. In addition, while up to half of patients with presumptive TB cannot produce adequate sputum specimens, current TB diagnostics rely on sputum-based tests. Therefore, the use of near point-of-care (nPOC) or point-of-care (POC) non-sputum-based tests can potentially provide more accessible TB diagnosis and reduce delays.

This CRCT is part of a larger series of studies within the EVIDENT Research Project in Indonesia. Based on a clinical validation study (EVIDENT work package 1) and a diagnostic yield, feasibility, and cost study (EVIDENT work package 2), the CRCT (EVIDENT work package 3) will provide evidence of the effects of implementation of a multi-component public health intervention in the intervention arm, compared to the control arm. Carefully designed clinical algorithms will be employed to incorporate the new diagnostic test, using sputum and/or tongue swab specimens, into the health services. To increase patients' attendance and utilisation of the new diagnostic test, a promotional package will be provided to clinics unable to host it and to selected pharmacies. Finally, a household contact investigation will be conducted, involving community health volunteers.

Clusters are the community health centre (CHC) catchment areas, defined as geographical areas surrounding a CHC where the TB programme is expected to be implemented. The interventions will be administered in HCFs and the community in the intervention arm, while the control arm will continue standard of care with no intervention, except for refresher training on TB case notification into the National TB Information System (locally known as Sistem Informasi Tuberkulosis or SITB) before the intervention roll-out. The primary and secondary endpoints will be assessed over the 12-month post-intervention roll-out (follow-up period), with adjustment for baseline (12-month pre-randomisation period). TB case notification data will be obtained from the National TB Information System.

In addition to the main study, several sub-studies will be conducted to assess the secondary objectives: the Patient Pathway & Patient Costing Sub-study, the Standardised Patient Sub-study, and the Health System Costing Sub-study. The Patient Pathway & Patient Costing study is a cross-sectional study of patients recently diagnosed with TB at the selected HCF in the intervention and control arms. In the Standardised Patient Sub-study, trained standardised patients will visit selected HCFs to present a clinical scenario and record their experiences regarding examinations, diagnostic testing, and referrals. The health system costing study will gather information on the costs of diagnosing TB in HCFs and communities in the intervention and control arms.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between >28 days and 14 years old with the following symptoms:

   * Cough ≥2 weeks
   * Acute malnutrition
   * Weight loss or weight faltering during the past 3 months among those who had contact history with patients with TB in the past 12 months.
2. Aged ≥15 years old who had a cough for ≥2 weeks or bloody cough, with or without the following symptoms:

   * Cough with/without sputum
   * Fever
   * Weight loss
   * Night sweat
   * Fatigue
   * Chest pain/discomfort
   * Breathlessness
   * Loss of appetite
   * Shivering

Exclusion Criteria:

* Have started TB treatment or TB prophylaxis therapy.

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in TB case notifications per population attending healthcare facilities | The outcome is measured for the 12 months before the commencement of any study procedures and over the 12-month follow-up period, starting 6 months after the start of the intervention roll-out.
  Difference in average TB notification rate per population attending healthcare facilities in intervention and control arms.

SECONDARY OUTCOMES:
Change in TB case notifications in CHC areas, who live in the area, per CHC area population | The outcome is measured for the 12 months before the commencement of any study procedures and over the 12-month follow-up period, starting 6 months after the start of the intervention roll-out.
  Difference in average TB notification rate among those who live in the CHC area, per CHC area population, in the intervention and control arms.
Change in proportion of microbiologically confirmed TB cases over all diagnosed TB cases | The outcome is measured over the 12 months before the commencement of any study procedures and over a 12-month follow-up period starting 6 months after the start of intervention roll-out.
  The proportion of microbiologically confirmed TB cases among all diagnosed cases in healthcare facilities in the intervention and control arms.
Difference in time to TB diagnosis from the beginning of symptoms (Patient Pathway and Patient Costing Sub-study) | Up to 10 months during the follow-up period
  The mean difference in days from symptom onset to TB diagnosis between the intervention and control arms.
Difference in time to TB diagnosis from the first visit to a formal HCF (Patient Pathway and Patient Costing Sub-study) | Up to 10 months during the follow-up period.
  The mean difference in days from the first visit to a formal HCF to TB diagnosis between the intervention and control arms.
Number of visits to healthcare facilities before TB diagnosis (Patient Pathway and Patient Costing Sub-study) | Up to 10 months during the follow-up period.
  Ratio of the mean number of visits to HCF before TB diagnosis among patients with TB notified in the intervention arm to that in the control arm.
Propensity to test for TB (Standardised Patient Sub-study) | Up to 6 months during the follow-up period
  Odds ratio comparing the odds of a standardised patient visit correctly resulting in a test for TB in the intervention and control arms.
Patient costs for TB diagnosis (Patient Pathway and Patient Cost Sub-study) | Up to 10 months during the follow-up period.
  Patient costs include medical and non-medical costs. Patient cost data will be collected from patients with TB diagnosed at CHCs, clinics, or hospitals. The patient cost data will be grouped into those diagnosed in the intervention and control arms.
TB diagnostic costs in the healthcare facilities and community settings (Health System Costing Sub-study) | Up to 6 months during the follow-up period.
  Health system costs will include building, equipment, supplies, training, and salary costs associated with TB diagnosis in the HCFs and community settings. Each cost will be grouped based on the intervention and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Bachti Alisjahbana, Professor, MD, PhD, Principal Investigator — Research Center for Care and Control of Infectious Diseases Universitas Padjadjaran
Locations (1):
- Bandung District Health Office, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
This CRCT aims to evaluate the effect of the diagnostic intervention package at the cluster level, including context-specific clinical algorithms that may greatly vary from those in other settings. The primary study outcomes will also be reported at the cluster level.

REFERENCES:
- [Background] Lestari BW, McAllister S, Hadisoemarto PF, Afifah N, Jani ID, Murray M, van Crevel R, Hill PC, Alisjahbana B. Patient pathways and delays to diagnosis and treatment of tuberculosis in an urban setting in Indonesia. Lancet Reg Health West Pac. 2020 Nov 28;5:100059. doi: 10.1016/j.lanwpc.2020.100059. eCollection 2020 Dec. PMID 34327397
- [Background] Sakundarno M, Nurjazuli N, Jati SP, Sariningdyah R, Purwadi S, Alisjahbana B, van der Werf MJ. Insufficient quality of sputum submitted for tuberculosis diagnosis and associated factors, in Klaten district, Indonesia. BMC Pulm Med. 2009 May 8;9:16. doi: 10.1186/1471-2466-9-16. PMID 19426477
- [Background] Pai M, Dewan PK, Swaminathan S. Transforming tuberculosis diagnosis. Nat Microbiol. 2023 May;8(5):756-759. doi: 10.1038/s41564-023-01365-3. No abstract available. PMID 37127703
- [Background] Church EC, Steingart KR, Cangelosi GA, Ruhwald M, Kohli M, Shapiro AE. Oral swabs with a rapid molecular diagnostic test for pulmonary tuberculosis in adults and children: a systematic review. Lancet Glob Health. 2024 Jan;12(1):e45-e54. doi: 10.1016/S2214-109X(23)00469-2. PMID 38097297
- [Background] Steadman A, Andama A, Ball A, Mukwatamundu J, Khimani K, Mochizuki T, Asege L, Bukirwa A, Kato JB, Katumba D, Kisakye E, Mangeni W, Mwebe S, Nakaye M, Nassuna I, Nyawere J, Nakaweesa A, Cook C, Phillips P, Nalugwa T, Bachman CM, Semitala FC, Weigl BH, Connelly J, Worodria W, Cattamanchi A. New Manual Quantitative Polymerase Chain Reaction Assay Validated on Tongue Swabs Collected and Processed in Uganda Shows Sensitivity That Rivals Sputum-based Molecular Tuberculosis Diagnostics. Clin Infect Dis. 2024 May 15;78(5):1313-1320. doi: 10.1093/cid/ciae041. PMID 38306491
- See also: EVIDENT Indonesia Official Website — https://evident.rc3id.unpad.ac.id/